CLINICAL TRIAL: NCT07249736
Title: "KETOMED: Ketonemia and Emergence Delirium in Children Undergoing General Anesthesia - A Multicenter Observational Study"
Brief Title: "KETOMED: Ketonemia and Risk of Emergence Delirium in Children Undergoing General Anesthesia - A Multicenter Observational Study"
Acronym: KETOMED
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Eva Lopez Santin, Investigator, Pediatric Anesthesia Department, Hospital Clínico Universitario de Valladolid, Hospital Clínico Universitario de Valladolid
Other Study IDs: Unique Protocol ID: PI-GR-25-4
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Emergence Delirium in Pediatric Anesthesia; Perioperative Ketonemia and Its Association With Recovery Outcomes in Children
Keywords: Pediatric anesthesia; Emergence delirium; Ketonemia; Perioperative monitoring; Multicenter observational study
MeSH Terms: conditions — Emergence Delirium; Ketosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for ketone measurement (serum or whole blood) collected perioperatively.
  Samples will be stored temporarily for ketone analysis and then discarded according to standard laboratory procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Anesthesia Cohort: This cohort includes children undergoing elective general anesthesia at participating centers. Participants will receive standard clinical care without experimental interventions. Blood samples will be collected perioperatively to measure ketone levels, and emergence delirium will be monitored using validated scales. Clinical and demographic data will also be recorded to explore potential risk factors associated with emergence delirium.

SUMMARY:
The objective of this observational study is to evaluate the relationship between ketonemia and emergence delirium in children undergoing general anesthesia. The main questions it aims to answer are:

* Does the level of ketonemia correlate with the risk of emergence delirium in pediatric patients?
* Are there specific perioperative factors that influence this relationship?

If there is a comparison group: Not applicable, as this is an observational study without intervention groups.

Participants will be asked to:

* Provide clinical and demographic information relevant to anesthesia and perioperative care.
* Undergo standard perioperative monitoring, including ketonemia measurement.
* Allow researchers to record anesthesia and recovery outcomes related to emergence delirium.

DETAILED DESCRIPTION:
KETOMED is a multicenter observational study designed to investigate the relationship between ketonemia and emergence delirium in pediatric patients undergoing general anesthesia. The study will prospectively collect perioperative data from children aged 2 to 12 years who are scheduled for elective procedures under general anesthesia.

Blood ketone levels will be measured at standardized time points during the perioperative period, and patients will be monitored for signs of emergence delirium using validated scales (e.g., Pediatric Anesthesia Emergence Delirium scale). In addition to ketonemia, perioperative variables such as type of anesthetic agents, duration of anesthesia, fasting status, and demographic information will be recorded to identify potential confounding factors.

The study aims to characterize the incidence of emergence delirium in relation to ketone levels and to explore whether specific metabolic or perioperative conditions are associated with higher risk. No experimental interventions will be applied; all patients will receive standard clinical care. The study is multicenter, allowing collection of data across diverse pediatric populations and surgical procedures, enhancing generalizability.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 12 years
* Elective procedure under general anesthesia
* Inpatient or Ambulatory Surgery Center (ASC) setting

Exclusion Criteria:

* Age younger than 2 years or older than 12 years
* Emergency surgery
* Postoperative admission to the Pediatric Intensive Care Unit (PICU)
* Neuropsychiatric disorder
* Carbohydrate metabolism disorder
* Declines to participate voluntarily in the study

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population includes children aged 2 to 12 years undergoing elective procedures under general anesthesia at participating centers. Participants may be admitted as inpatients or treated in an Ambulatory Surgery Center (ASC). Children with neuropsychiatric disorders, carbohydrate metabolism disorders, those undergoing emergency surgery, or requiring postoperative admission to the Pediatric Intensive Care Unit (PICU) are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Emergence Delirium in Pediatric Patients | During the immediate postoperative recovery period (typically 30-60 minutes after emergence from anesthesia)
  The proportion of children experiencing emergence delirium during the recovery period after general anesthesia, assessed using a validated scale (e.g., Pediatric Anesthesia Emergence Delirium scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided